CLINICAL TRIAL: NCT02817308
Title: Correlation of Serum CA19-9 Levels With Levels in Saliva and Urine of Patients With Ductal Adenocarcinoma of the Pancreas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CA19-90415-15-RMBCTIL
Record Dates: First submitted 2016-02-10; First posted 2016-06-29 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Carcinoma, Pancreatic Ductal
Keywords: Antigen, CA-19-9; Salivas; body fluids
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal | interventions — Urination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients (Experimental): Patients with a proven diagnosis of ductal adenocarcinoma of the pancreas with elevated levels of CA19-9 and possibly elevated CEA levels.
  intervention: samples of blood, saliva and urine
  Interventions: Other: samples of blood, saliva and urine
- Control (Other): Patients or healthy volunteers with out a known evidence of malignancy with presumably normal levels of CA19-9 and CEA.
  intervention: samples of blood, saliva and urine
  Interventions: Other: samples of blood, saliva and urine

INTERVENTIONS:
Other: samples of blood, saliva and urine — Spot samples of Blood, urine and saliva

SUMMARY:
Ductal adenocarcinoma of the pancreas is the fifth leading cause of cancer related deaths in the European Union. Tumor markers CA19-9 and carcinoembryonic antigen are important components in decision making and follow-up of patients diagnosed with this disease.

These tumor markers were found to be elevated not only in the serum but also in other body fluids in patients with malignant lesions of the parotid gland and the urinary tract. The authors have described in a previews small preliminary study a positive and a strong linear correlation between the levels of CA19-9 in urine and saliva with those presented in the serum of patients with ductal adenocarcinoma of the pancreas. The current study seeks to enlarge the study population to confirm the previous results and standardize the measured levels of CA19-9 in these body fluids.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Proven diagnosis of ductal adenocarcinoma of the pancreas
* elevated levels of CA19-9
* possible elevated levels of CEA

Exclusion Criteria:

Controls:

* Previous diagnosis of malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-07; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
correlation of CA19-9 levels in urine and saliva with those in the serum | 1 year

SECONDARY OUTCOMES:
Number of participants needed to standardize the measurements in urine and saliva according to those measured in the serum. | 1 year
  upper and lower levels of CA19-9 measured in urine and saliva are not yet standardized. and repeated measurements in these body fluids compared to the ones in serum of healthy subjects are needed for such standardization.

CONTACTS AND LOCATIONS:
Overall Officials: Offir Ben-Ishay, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam - health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No